CLINICAL TRIAL: NCT02784379
Title: The Comparison Both of the Electromyography Results of the Pectoral Muscle in Unilateral Mastalgia Patients
Brief Title: Electromyography of the Pectoral Muscle in Mastalgia Patients
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, M.D., Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: Mastalgia
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Mastalgia
Keywords: Mastalgia; electromyography; Pectoral
MeSH Terms: conditions — Mastodynia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- The breast with mastalgia: Electromyography will be performed to the pectoral muscle that is placed behind the breast with mastalgia.
- The breast without mastalgia: Electromyography will be performed to the pectoral muscle that is placed behind the breast without mastalgia.

SUMMARY:
Mastalgia is a common problem for women. The aim of this study is to investigate the role of neuromuscular pathologies of the thorax wall at mastalgia ethiopathogenesis.

DETAILED DESCRIPTION:
Mastalgia is a common health problem for women especially these days. Studies demonstrated that 48% of the women with mastalgia have serious difficulties in their sexual life, 36% have physical activity difficulties, 13% have social activity difficulties and 6% have work or school activity difficulties. The etiology of the mastalgia is not clear. Because of the women with mastalgia tested out lots of examinations for the etiology. Also this problem has financial load because of the unknown etiology.

ELIGIBILITY:
Inclusion Criteria:

* Subject has unilateral mastalgia

Exclusion Criteria:

* Subject has pregnancy
* Subject has breast cancer
* Subject has a history of breast operation
* Subject has diabetes mellitus
* Subject has 1 cm or above cystic or solid lesions in the breasts.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 31 patients who has unilateral mastalgia
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Electromyography results of the pectoral muscle. | 5 days
  The electromyography results of the pectoral muscle which are placed behind the healthy breast (group 1) and the breast with mastalgia (group 2) will be evaluated. The results of the both groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Cemal Kaya, M.D., Principal Investigator — Sisli Etfal Training and Research Hospital
Locations (1):
- Sisli Etfal Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kernerman E, Park E. Severe Breast Pain Resolved with Pectoral Muscle Massage. J Hum Lact. 2014 Aug;30(3):287-291. doi: 10.1177/0890334414535842. Epub 2014 May 29. PMID 24874898
- [Result] Joyce DP, Alamiri J, Lowery AJ, Downey E, Ahmed A, McLaughlin R, Hill AD. Breast clinic referrals: can mastalgia be managed in primary care? Ir J Med Sci. 2014 Dec;183(4):639-42. doi: 10.1007/s11845-013-1066-z. Epub 2014 Jan 9. PMID 24402166
- [Result] Salzman B, Fleegle S, Tully AS. Common breast problems. Am Fam Physician. 2012 Aug 15;86(4):343-9. PMID 22963023